CLINICAL TRIAL: NCT06850948
Title: Exploring the Experiences of Gender Identity Healthcare for Autistic Transgender/ Gender Diverse Adults
Brief Title: Experiences of Healthcare for Autistic TGD Adults
Status: Not yet recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 25003
Record Dates: First submitted 2025-02-26; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Autism Spectrum Disorder (ASD
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Evaluation Studies as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Qualitative — Interviews collected with participants concerning their experience of gender identity healthcare

SUMMARY:
To explore the experiences of autistic gender diverse adults that have attempted or are attempting to access, have accessed or are currently accessing gender identity healthcare in the United Kingdom

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years or older, they must have first-hand experiences of currently accessing, previously having accessed, or having attempted to access NHS Gender identity clinics in the United Kingdom. The participant must identify as TGD in some capacity (e.g. transgender, nonbinary) and have a formal diagnosis of autism. (Proof of formal diagnosis will not be sought, but participants will be asked about information on this. Diagnosis of autism be asked on the demographic questionnaire, along with question on the diagnosis procedure (e.g. service diagnosis, age of diagnosis). The participant must be able to communicate (verbal or written) in the English Language and be able to provide informed consent.

Exclusion Criteria:

* People who do not meet the inclusion criteria will be excluded from the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender, Non-binary, gender diverse and all that do not fall into the binary cisgender man or cisgender man
Study Population: The present study will be promoted via the NHS at the Nottingham Centre for Transgender Health, for which advertisements of the study (see attached document) will be displayed within the clinic
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2025-03-03 (Estimated); Primary Completion 2026-09-07 (Estimated); Study Completion 2026-09-07 (Estimated)

PRIMARY OUTCOMES:
Interview | From March 2025 to September 2026
  Qualitative interview

IPD SHARING:
Plan to Share IPD: Undecided